CLINICAL TRIAL: NCT01527903
Title: Sedation of Surgical Patients in the Intensive Care Unit: A Randomized Comparison Between Propofol-Remifentanil and Midazolam-Remifentanil Sedation
Brief Title: A Comparison Between Propofol-Remifentanil and Midazolam-Remifentanil Sedation in the Intensive Care Unit
Acronym: ICU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2009-0311
Record Dates: First submitted 2012-01-24; First posted 2012-02-07 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Sedation
Keywords: propofol; midazolam; sedation; ICU

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propofol (Active Comparator)
  Interventions: Drug: Propofol infusion
- Midazolam (Active Comparator)
  Interventions: Drug: Midazolam infusion

INTERVENTIONS:
Drug: Propofol infusion — IV propofol 2% at a rate of 1.0 mg kg-1 h-1, increments or decrements of 0.1 mg kg-1 h-1
  Arms: Propofol
Drug: Midazolam infusion — midazolam at a rate of 0.1 mg kg-1 h-1, increments or decrements of 0.05 mg kg-1 h-1
  Arms: Midazolam

SUMMARY:
The purpose of this study is to compare propofol-remifentanil sedation with midazolam-remifentanil sedation in regards to extubation and weaning time, length of stay in the ICU, as well as the incidence of delirium. Primary end-points were weaning time and extubation time, and secondary end-points were the incidence of delirium and length of stay in the ICU.

DETAILED DESCRIPTION:
With on-going emphasis on early extubation, as well as further recognition of morbidity and mortality associated with delirium, the specific sedatives and analgesics used in the ICU is an issue of interest. Recent studies have focused on comparing sedatives, but interpretations are often confounded by the fact that in most studies, different analgesics were used when comparing two sedative medications. The role of remifentanil as the main analgesic in the ICU is being recognized. Pharmacodynamic and pharmacokinetic profiles of remifentanil makes it an ideal analgesic in the ICU setting. The investigators therefore designed this randomized study to compare sedation with propofol and midazolam in a remifentanil-based sedation and analgesia.

The purpose of this study is to compare propofol-remifentanil sedation with midazolam-remifentanil sedation in regards to extubation and weaning time, length of stay in the ICU, as well as the incidence of delirium. Primary end-points were weaning time and extubation time, and secondary end-points were the incidence of delirium and length of stay in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* surgical patients over 18 years old who were admitted to the ICU for postoperative ventilator care after sevoflurane-remifentanil based general anesthesia

Exclusion Criteria:

* pre-existing neurologic dysfunction (dementia)
* head trauma patients
* previous history of alcohol abuse or substance abuse
* patients who had baseline serum creatinin levels of over 2.5mg/100ml
* uncompensated liver cirrhosis
* hemorrhagic, cardiogenic, or septic shock
* pregnancy or breast feeding
* tracheostomy or extubation before ICU admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Extubation time | monitored from dicontinuation of sedatives to extubation, during an expected average of 3 hours
  the time to extubation : defined as the time from discontinuation of infusion to extubation

SECONDARY OUTCOMES:
delirium | monitored during the entire ICU stay (an expected average of 6 days)
  delirium assessed by Confusion Assessment Method for ICU (CAM-ICU)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea